CLINICAL TRIAL: NCT05420935
Title: Repertoire and Properties of Anti-drug Antibodies Involved in Immediate Hypersensitivity in the Operating Room
Acronym: MEDIREP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211277
Record Dates: First submitted 2022-05-20; First posted 2022-06-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypersensitivity, Immediate; Peri-operative Injury; Antibiotic Allergy; Antibody Hypersensitivity
Keywords: Hypersensitivity, IgE, IgG, repertoire, NMBA, anaphylaxis
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity; Epilepsy, Idiopathic Generalized; Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IgG group (Other): Patient in the IgG group will benefit from a blood sampling of 5 ml (for realization of a basophil activation test) and a blood sampling of 250 ml
  Interventions: Diagnostic Test: IgG group
- IgE group (Other): Patient in the IgE will benefit from a blood sampling of 5 ml (for realization of a basophil activation test) and a bone marrow sampling (approx 2 ml)
  Interventions: Diagnostic Test: IgE group
- IgG group + IgE group (Other): Patient in the IgG + IgE will benefit from a blood sampling of 5 ml (for realization of a basophil activation test), a blood sampling of 250 ml and a bone marrow sampling (approx 2 ml)
  Interventions: Diagnostic Test: IgG group + IgE group

INTERVENTIONS:
Diagnostic Test: IgG group — Will be performed :
  * a blood sampling of 5 ml (for realization of a basophil activation test)
  * a blood sampling of 250 ml
  Arms: IgG group
Diagnostic Test: IgE group — Will be performed :
  * a blood sampling of 5 ml (for realization of a basophil activation test)
  * a bone marrow sampling
  Arms: IgE group
Diagnostic Test: IgG group + IgE group — * a blood sampling of 5 ml (for realization of a basophil activation test)
  * a blood sampling of 250 ml
  * a bone marrow sampling
  Arms: IgG group + IgE group

SUMMARY:
Acute per-anesthetic hypersensitivity reaction (HSA-PA) is a rapidly occurring systemic reaction following injection of a drug during anesthesia (mortality between 3 and 9%). The substances responsible for these reactions in France are curare in 60% of cases, followed by antibiotics. The main mechanism mentioned is an immediate systemic hypersensitivity immune reaction mediated by IgE antibodies (anaphylaxis). NeuroMuscular Blocking Agents (NMBA; curare) relax skeletal muscles to facilitate surgeries and permit intubation, but lead to adverse reactions: (a) severe hypersensitivity reactions (anaphylaxis) thought to rely on pre-existing anti-NMBA antibodies; (b) complications due to postoperative residual curarization. Identification of patients at risk remains suboptimal due to the lack of adequate tools to detect anti-NMBA antibodies. A capturing agent exists for only one out of the four most used NMBAs, allowing reversal of profound curarization. Case reports suggested that it might also ameliorate an ongoing anaphylaxis due to that NMBA.

Based on strong preliminary results, our study proposes to characterize anti-drugs antibody repertoires in patients with various NMBA or antibiotics-anaphylaxis, describe activation pathways leading to anaphylaxis, develop and validate diagnostic and therapeutic molecules to ameliorate patient screening, NMBA-anaphylaxis and reverse profound neuromuscular block.

DETAILED DESCRIPTION:
Acute per-anesthetic hypersensitivity reaction (HSA-PA) is a rapidly occurring systemic reaction following injection of a drug during anesthesia (mortality between 3 and 9%). The substances responsible for these reactions in France are curare in 60% of cases, followed by antibiotics. The main mechanism mentioned is an immediate systemic hypersensitivity immune reaction mediated by IgE antibodies (anaphylaxis).

NeuroMuscular Blocking Agents (NMBA; curare) used in the clinic (e.g., atracurium, suxamethonium, rocuronium, vecuronium) belong to the curare family and block the nicotinic acetylcholine receptor to cause muscle relaxation. They share the presence of quaternary ammonium groups that are required for binding the acetylcholine receptor, and thus for their biological activity. Even though NMBA are relatively safe molecules, two main types of adverse reactions have been reported.

The most striking are immediate and severe anti-drug reactions at NMBA infusion with 1/10,000 patients suffering from severe hypersensitivity reactions, i.e. anaphylaxis. Anaphylaxis is classically considered to rely on IgE antibodies against the culprit compound, and to involve massive histamine liberation by mast cells and basophils, following antigen-induced aggregation of IgE receptor (FcεRI)-bound specific IgE antibodies1. The clinical diagnosis of anaphylaxis to NMBA is based on this IgE paradigm. NMBA quaternary ammonium cations are considered their major allergenic epitopes2, even if patients are rarely hypersensitive to several NMBA, even closely related NMBA like rocuronium and vecuronium that derive from each other, suggesting that antibodies may bind NMBA-specific structures other than quaternary ammoniums. Antibodies may even interact with NMBA as a "whole" epitope due to NMBA very reduced size; NMBA indeed vary from 300-1,000 Da. Intriguingly, 10-20% of patients who experience NMBA-induced anaphylaxis do not present with any biological signs of IgE-dependent immune activation, suggestive of other potential mechanisms. 4 An IgG antibody pathway has recently been described in NMBA-induced human anaphylaxis, leading to Platelet-Activating Factor release, neutrophil and platelet activation, which may aggravate anaphylaxis in combination with the IgE-pathway or underlie anaphylaxis in the absence of specific IgE.

The other most common adverse reaction is not allergic in nature, and is due to prolonged presence of NMBA following surgery, i.e. "residual curarization". This very frequent complication (up to 83% of the patients) leads to adverse postoperative pulmonary events, pharyngeal dysfunction, urgent tracheal reintubation and prolonged stay in post-anesthesia care units that lead to a high economic burden13. The first option for pharmacological neuromuscular blockade reversal, prostigmine (used for atracurium reversal), is restricted to situations where half of the spontaneous reversal is effective. The second one is a synthetic cyclodextrin, sugammadex, that captures rocuronium or vecuronium in vivo within minutes following injection. Instant blockade reversal might be necessary, as in difficult intubation scenarios, explaining that it has been considered economically advantageous to administer sugammadex despite a cost of $100/dose, leading to a $400-$3,000 economy per patient.

Based on strong preliminary results, our study proposes to characterize anti-drugs antibody repertoires in patients with various NMBA or antibiotics-anaphylaxis, describe activation pathways leading to anaphylaxis, develop and validate diagnostic and therapeutic molecules to ameliorate patient screening, NMBA-anaphylaxis and reverse profound neuromuscular block.

ELIGIBILITY:
Inclusion Criteria:

Common to both groups:

* Age ≥ 18 years old and ≤ 70 years old
* Patient having presented an allergic reaction in the operating room in the last 10 years, regardless of the grade of severity, the causative agent or the type of anesthesia
* Patient having benefited from an allergy-anaesthesia consultation in the investigator center

For IgE group:

- presence of at least one positive skin test to one of the suspected agent (curare and/or antibiotic) during the allergist consultation

For the IgG group:

- presence of circulating IgG-type antibodies directed against one of the suspected agents (curare, antibiotic, antiseptic), identified in the routine biological tests carried out at the time of the shock and / or the consultation of allergology.

Exclusion Criteria:

Common to both groups:

* Absence of written informed consent
* Protected person: under guardianship or curatorship
* Patient without social security
* Pregnancy of breast feeding
* Ongoing immunosuppressive or chemotherapy
* Acute heart failure
* Patient included in another interventional research with an exclusion period

For IgE group:

* Taking oral or injectable anticoagulants
* Taking a double antiplatelet aggregation
* Previous sternotomy
* Previous thoracic radiation therapy
* Known allergy to local anesthesic or iodinated skin products
* Previous major sternal cutaneous lesions

Prerequisites for carrying out the sternal sample in order to carry out a myelogram (IgE group):

* Leukocytes > 4 giga/L in the 2 months preceding inclusion
* Platelets > 100,000 / mm3 in the 2 months preceding inclusion

For the IgG group

* Orthostatic hypotension
* Realization of a blood donation in the 6 to 8 weeks preceding inclusion

Prerequisites for performing the blood sample (IgG group):

- Hemoglobin > 12.5 g/dL for women and > 13 g/dL for men in the 2 months preceding inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2033-04-12 (Estimated); Study Completion 2033-12-15 (Estimated)

PRIMARY OUTCOMES:
Obtain sequences of gene producers (VH and VL pairs) coding for the variable part of anti-drug antibodies, thanks to the isolation of B lymphocytes of antibodies directed against the responsible molecule, from blood cells or bone marrow | up to 10 years

SECONDARY OUTCOMES:
Production of recombinant antibodies based on obtained sequences | up to 10 years
  Purification system (AKTA 25L, Cytiva)
Evaluate antibodies properties, such as specificity | up to 10 years
  ELISA
Evaluate antibodies properties, such as avidity | up to 10 years
  Interferometry (Octet, ForteBio)
Ability of antibodies expressed as N297A mutated human IgG1 to reduce or block target curare-induced neuromuscular blockade without an immune response triggered by the antibody drug | up to 10 years
  Measure of muscle strength of mice
Ability of antibodies expressed as N297A mutated human IgG1 to reduce or block target curare-induced neuromuscular blockade without an immune response triggered by the antibody drug | up to 10 years
  Measure of motricity of mice
Ability of antibodies expressed as N297A mutated human IgG1 to reduce or block target curare-induced neuromuscular blockade without an immune response triggered by the antibody drug | up to 10 years
  Measure the survival rate of mice
Ability of antibodies expressed as N297A mutated human IgG1 to reduce or block target curare-induced neuromuscular blockade without an immune response triggered by the antibody drug | up to 10 years
  Evaluate the absence of occurrence of anaphylactic shock
Core temperature loss greater than 3°C within 60 minutes after target drug injection only in mice pre-injected with anti-drug IgE or IgG | up to 10 years
  Rectal probe thermometer for mice

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie Gouel, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat claude Bernard, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No